CLINICAL TRIAL: NCT06610552
Title: Real-life Implementation Randomized Clinical Trial Assessing Effectiveness of Powerly - Science-based Digital Intervention Preventing Postpartum Depression and Anxiety
Brief Title: Powerly - Science-based Digital Intervention Preventing Postpartum Depression and Anxiety
Acronym: POWERLY app
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marta Marciniak (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Marta Marciniak, Dr, Erasmus University Rotterdam
Organization: Erasmus University Rotterdam (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UZH24.08.23
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Stress; Postpartum Depressive Disorder; Postpartum Anxiety
Keywords: pregnancy; postpartum depression; postpartum anxiety; stress; digital health; mobile health; ecological momentary intervention
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Powerly (Experimental): Participants in the intervention group will complete baseline questionnaires and receive instructions on how to download Powerly. They will use the app daily for 28 days, at least once per day, and will be invited to complete the questionnaires again, and once more six weeks postpartum.
  Interventions: Behavioral: Powerly
- Care as usual (No Intervention): Participants in the CAU group will complete baseline questionnaires and be informed that they will receive access to Powerly six weeks postpartum. They will be invited to complete the questionnaires again 28 days later, and once more six weeks postpartum.

INTERVENTIONS:
Behavioral: Powerly — Powerly is a mental well-being mobile app, in which pregnant women can track their mood and level of stress, and receive personalized psychological modules to increase their mental health and well-being. By integrating evidence-based content and cognitive behavioral techniques with insights from pregnant and postpartum individuals and health professionals, Powerly offers a comprehensive psychological support including reappraisal, mental imagery, gratitude, mindfulness, self-efficacy and behavioral activation exercises.
  Arms: Intervention - Powerly

SUMMARY:
The goal of this clinical trial is to determine if the Powerly app can help prevent postpartum depression and anxiety in healthy pregnant women.

The main questions it aims to answer are:

* Does the Powerly app reduce postpartum depression and anxiety?
* Does it improve emotion regulation and maternal bonding with a child?

Researchers will compare two groups: one using the Powerly app and the other receiving care as usual (CAU) to see if the app leads to better mental health outcomes.

Participants will:

* Use the Powerly app for four weeks (if in the intervention group).
* Complete mental health assessments before the study, after four weeks, and six weeks postpartum.

DETAILED DESCRIPTION:
Pregnancy is a period of significant emotional and physical changes, with up to 30% of expecting mothers experiencing high stress. After birth, around 15-20% of new mothers suffer from postpartum depression, and 25-35% experience anxiety. Despite broad availability of mobile apps aimed at these challenges, none of them have been rigorously tested through clinical studies. To fill this gap, we developed Powerly, a science-based mobile app designed to help prevent postpartum depression and anxiety.

In this study, 140 healthy pregnant women will be randomly assigned to one of two groups: one will use the Powerly app for four weeks, while the other will receive care as usual (CAU). Powerly is grounded in cognitive behavioral therapy (CBT) and personalized to the individual's needs, with input from healthcare professionals and pregnant women. We will collect information on participants' mental health at three points: before they start using the app, after four weeks of app use / CAU, and six weeks after giving birth. The app's effectiveness will be evaluated by examining improvements in mental health outcomes, such as reduced rates of postpartum depression and anxiety, better emotion regulation, and stronger maternal bonding with a baby.

ELIGIBILITY:
Inclusion Criteria:

* being between 24 and 32 weeks pregnant,
* owning an iPhone,
* having sufficient fluency in German language

Exclusion Criteria:

* high-risk pregnancies,
* history of substance abuse and psychiatric disorders such as bipolar disorder, schizophrenia, or other psychotic disorders,
* current use of professional face-to-face psychotherapeutic support,
* participation in other clinical trials or interventions at the same time

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
DASS (Depression, Anxiety, and Stress Scales) | From baseline measurement until the second follow-up measurement at 6 weeks postpartum
  a validated set of brief scales consisting of 21 items used to measure the severity of depression, anxiety, and stress symptoms
PDSS (Postpartum Depression Screening Scale) | Collected only at second follow-up measurement 6 weeks postpartum
  a comprehensive tool comprising 35 items designed to identify symptoms of postpartum depression, including aspects such as sleep and eating disturbances, insecurity, emotional lability, guilt, and shame

SECONDARY OUTCOMES:
CERQ (Cognitive Emotion Regulation Questionnaire) | From baseline measurement until the second follow-up measurement at 6 weeks postpartum
  it comprises 36 items assessing the strategies individuals employ to manage their emotions, including positive reappraisal, acceptance, rumination, and putting into perspective, among others
PASS-C (Positive Appraisal Style scale - content) | From baseline measurement until the second follow-up measurement at 6 weeks postpartum
  comprises of 14 items and measures person's general style of evaluating stressors
BRS (Brief Resilience Scale) | From baseline measurement until the second follow-up measurement at 6 weeks postpartum
  it measures resilience operationalized as an outcome of the process of adaptation to adversity, using 5 questions
BSS-RI (Birth Satisfaction Scale - Revised Indicator) | Collected only at second follow-up measurement 6 weeks postpartum
  assesses the subjective experience of labor, including aspects of anxiety, stress, feelings of control, and support, using 6 items
PBQ (Postpartum Bonding Scale) | Collected only at second follow-up measurement 6 weeks postpartum
  the 25-item questionnaire measures the quality of the bond between the mother and her infant. It includes factors such as the general bonding factor, anxiety about the baby, and rejection
mARM (mobile Agnew Relationship Measure) | Collected only at first follow-up measurement after 4 weeks of study
  it evaluates the therapeutic alliance between the app and the user through 25 items. It covers topics such as confidence, openness, user initiative, and partnership
uMARS (user version of the Mobile Application Rating Scale) | Collected only at first follow-up measurement after 4 weeks of study
  tool used for assessment of the feasibility of the app, including aspects of engagement, aesthetics, functionality, and the quality of information provided in the EMI, with 20 questions
MFA (Maternal-Fetal Attachment Scale) | From baseline measurement until first follow-up measurement after 4 weeks of study
  the 24-item scale evaluates the bond between mother and fetus during pregnancy. It includes questions about interactions with the fetus, attributing characteristics to the fetus, and role-taking, among others
GSE (General Self-Efficacy Scale) | From baseline measurement until the second follow-up measurement at 6 weeks postpartum
  it evaluates an individual optimistic self-belief in their capability to handle difficult tasks, challenges, and adversities, through 10 items
Adherence | Collected passively during app use period (4 weeks)
  the number of interactions with the app by each of the participants

OTHER OUTCOMES:
BFI-10 (Big Five Inventory-10) | Collected only during baseline measurement
  it assesses the five major dimensions of personality (openness, conscientiousness, extraversion, agreeableness, and neuroticism) with 10 items
PMH (Positive Mental Health scale) | Collected only during baseline measurement
  includes nine items to measure specifically positive mental well-being

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Anonymized questionnaire (self-report) data will be shared in an open science repository, for instance Open Science Framework.
Supporting Information: Study Protocol
Time Frame: The data will be shared after the study completion (published along with manuscripts from the trial), without the end date.
Access Criteria: The data will be publicly available.

REFERENCES:
- [Derived] Marciniak MA, Rohde J, Yuen KSL, Binder H, Walter H, Wieser MJ, Kalisch R, Roelofs K, Kleim B. Development of Powerly, unguided mobile app intervention preventing postpartum depression and anxiety & study protocol of randomized clinical trial. Internet Interv. 2025 Jun 16;41:100843. doi: 10.1016/j.invent.2025.100843. eCollection 2025 Sep. PMID 40607107